CLINICAL TRIAL: NCT03109379
Title: A Prospective, Multi-center, Open-label Study of Trospium Delivered Intravesically by TAR-302-5018 to Subjects With Idiopathic Overactive Bladder (iOAB) and Urinary Incontinence
Brief Title: Safety and Tolerability of TAR-302-5018 in Subjects With Idiopathic Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taris Biomedical LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAR-302-103
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Overactive Bladder With Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAR-302-5018 (42-day Indwelling) (Experimental): Trospium-Releasing Intravesical System (TAR-302-5018) is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 42. TAR-302-5018 releases trospium gradually during the 42 day indwelling time.
  Interventions: Drug: Trospium-Releasing Intravesical System (TAR-302-5018)
- TAR-302-5018 (84-day Indwelling) (Experimental): Trospium-Releasing Intravesical System (TAR-302-5018) is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 84. TAR-302-5018 releases trospium gradually during the 84 day indwelling time.
  Interventions: Drug: Trospium-Releasing Intravesical System (TAR-302-5018)

INTERVENTIONS:
Drug: Trospium-Releasing Intravesical System (TAR-302-5018) — TAR-302-5018 is a passive, nonresorbable trospium-releasing intravesical system whose primary mode of action is the controlled release of trospium into the bladder over a 42-day period.

SUMMARY:
The purpose of this study is to determine if TAR-302-5018, an investigational drug-delivery system, is safe and tolerable in patients with idiopathic overactive bladder and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria (Part 1):

1. Symptoms of overactive bladder (OAB) (frequency/urgency) with urge urinary incontinence or mixed urinary incontinence with a predominant urge component for at least 6 months

   * 8 or more voids per 24 hours as recorded in a diary
   * At least 4 incontinence episodes associated with urgency recorded in a 3-day diary.

     * At least 1 episode must occur per each 24 hour day
2. Inadequate response or limiting side effects with anticholinergics for the treatment of OAB

Exclusion Criteria (Part 1):

1. Age <18 years.
2. OAB caused by neurological condition.
3. Presence of significant renal dysfunction at screening (Glomerular Filtration Rate <30 mL/min).
4. Presence of significant polyuria of any cause at screening (urine output >4,000 mL/day).
5. History of pelvic radiation.
6. History of either bladder cancer or bladder pathology that the investigator deems unfit for study inclusion.
7. Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome.
8. Subjects with any bladder or urethral anatomic feature that may prevent the safe placement, indwelling use, or removal of TAR 302 5018.
9. In the opinion of the investigator, the subject has a history of significant stress urinary incontinence.
10. Subjects with active bladder stones or history of bladder stones <6 months prior to study entry.
11. History of recurrent symptomatic urinary tract infections (UTIs) (>4 per 1 year).
12. Subjects with either urinary retention or gastric retention or uncontrolled narrow-angle glaucoma.
13. A post-void residual volume (PVR) of 300 mL or greater
14. Subjects with known hypersensitivity to trospium, chemically-related drugs, or component excipients.
15. Subjects with known hypersensitivity to the device materials, including silicone and nitinol.
16. Subjects actively taking oral trospium.
17. The addition of a new or a change in dose to a current medication for the treatment of OAB (i.e. anticholinergics, beta-3 adrenergic agonists, antispasmodics, antidepressants, or hormones) within 30 days prior to signing the informed consent form (ICF). A stable dose must continue through the final study visit. If previously used and discontinued, these medications must have been stopped for >2 weeks prior to Day 0.
18. Intravesical onabotulinum toxin use within the last 9 months prior to the Screening Visit.
19. Intravesical anticholinergic medications within the last 30 days prior to the Screening Visit.
20. History of non-medication based therapy (i.e. InterStim therapy) for the treatment of OAB. History of non-invasive neuromodulation (i.e. Percutaneous Tibial Nerve Stimulation (PTNS)) is allowed if discontinued at least 8 weeks prior to Study Day 0.
21. Female subject who is pregnant (as verified by urine test at time of screening) or lactating or of childbearing potential and not using acceptable methods of contraception.
22. Subject has a medical condition that may cause noncompliance with the study protocol.
23. Subject refuses to provide written informed consent.
24. Subject will be unable or unwilling to complete the questionnaires, diaries, or attend all protocol mandated study visits.
25. Participation in another drug, device, or behavioral study within 60 days prior to the Screening Visit.
26. History or presence of any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, gynecological, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder that, in the opinion of the investigator, contraindicates participation.
27. History of any of the following within 3 months prior to Screening Visit:

    * Major illness/major surgery (requiring hospitalization), including pelvic, lower back surgery or procedure unrelated to bladder cancer; most outpatient procedures are not exclusionary
    * Renal or ureteral stone disease or instrumentation
    * Childbirth
28. Difficulty providing blood samples.
29. Other unspecified reasons that, in the opinion of the investigator or TARIS, make the subject unsuitable for enrollment.

Inclusion Criteria (Part 2):

1. Symptoms of idiopathic overactive bladder (iOAB) (frequency/urgency) with urge urinary incontinence or mixed urinary incontinence with a predominant urge component for at least 6 months.

   * 8 or more voids per 24 hours as recorded in a diary
   * At least 4 incontinence episodes associated with urgency recorded in a 3-day diary.

     1. At least 1 episode must occur per each 24 hour day
2. In the opinion of the investigator, the subject has experienced an inadequate response to or limiting side effects with prior oral medications for the treatment of OAB.

Exclusion Criteria (Part 2):

1. Age <18 years.
2. Neurologic bladder condition.
3. Subjects with Diabetes Mellitus (both Type 1 & Type 2) must demonstrate optimal glycemic control with HbA1c levels < 7.5 % and an absence of significant glucosuria defined as 3+ glucose via dipstick at screening.
4. Presence of significant polyuria of any cause at screening (urine output >3,000 mL/day).
5. Presence of nocturnal polyuria at time of study screening defined as >30% of total 24-hour urine collected from time of evening (P.M.) sleep and inclusive of the first morning (A.M.) void.
6. History of pelvic irradiation.
7. History of either bladder cancer or bladder pathology that the investigator deems unfit for study inclusion.
8. Currently uses intermittent catheterization (IC) to empty the bladder within 30 days of Day 0.
9. Subjects with any bladder or urethral anatomic feature (e.g., urethral stricture) that in the opinion of the investigator may prevent the safe placement, indwelling use, or removal of IP.
10. Subjects with active bladder stones or history of bladder stones < 6 months prior to study entry.
11. Gross hematuria within 30 days of Day 0.
12. History of uncontrolled bleeding, bleeding diathesis, or underlying coagulopathy within 30 days of Day 0.
13. In the opinion of the investigator, the subject has a history of predominance of significant stress urinary incontinence.
14. History of > 2 symptomatic urinary tract infections in the 6-months prior to Day 0.
15. Subjects with either urinary retention or gastric retention or uncontrolled narrow-angle glaucoma within 90 days of Day 0.
16. A post-void residual volume (PVR) of 100-mL or greater.
17. Subjects with known hypersensitivity to trospium, chemically-related drugs, or component excipients.
18. Subjects with known hypersensitivity to the device materials, including silicone and nitinol.
19. Anticholinergic or beta-3 agonist use for the treatment of urge urinary incontinence < 2 weeks prior to Day 0.
20. History of intravesical onabotulinum toxin use within the last 9 months prior to the Screening Visit.
21. Intravesical anticholinergic medications within the last 14 days prior to the Screening Visit.
22. History of procedural-based neuromodulation therapy (e.g. InterStim therapy, Percutaneous Tibial Nerve Stimulation [PTNS]) for the treatment of OAB.
23. Female subject who is pregnant (as verified by serum test at time of screening) or lactating.
24. Subject has, in the opinion of the investigator, a medical condition that may cause noncompliance with the study protocol.
25. Subject who is unable or unwilling to complete the questionnaires, diaries, or attend all protocol mandated study visits.
26. Participation in another drug, device, or behavioral study within 60 days prior to the Screening Visit.
27. History or presence of any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, gynecological, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder, or other unspecified reasons that, in the opinion of the investigator or TARIS, make the subject unsuitable for enrollment.
28. History of any of the following within 3 months prior to Screening Visit:

    i. Major illness/major surgery (requiring hospitalization), including pelvic, lower back surgery or procedure; most outpatient procedures are not exclusionary.

    ii. Childbirth.
29. History of prostatic biopsy or surgery (ablative or non-ablative) within 6 months prior to Day 0.
30. History of significant pelvic organ prolapse (Grade >/= 3).
31. Difficulty providing blood samples.
32. Known history of drug or alcohol dependency within 12 months of screening.
33. Other unspecified reasons that, in the opinion of the investigator or TARIS, make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Safety of TAR-302-5018 assessed throughout the study based on reported AEs (Part 1) | Upon insertion, 42-day continuous exposure, and removal
  Safety will be assessed throughout the study based on reported AEs, investigational product events (IPEs), physical examinations (PEs), vital signs, clinical laboratory tests, scheduled cystoscopic examinations, bladder ultrasounds, bladder post-void residual volume (PVR), and the use of concomitant medications.
Safety of TAR-302-5018 assessed throughout the study based on reported AEs (Part 2) | Upon insertion, 84-day continuous exposure, and removal
  Safety will be assessed throughout the study based on reported AEs, investigational product events (IPEs), physical examinations (PEs), vital signs, clinical laboratory tests, scheduled cystoscopic examinations, bladder ultrasounds, bladder post-void residual volume (PVR), and the use of concomitant medications.

SECONDARY OUTCOMES:
Tolerability of TAR-302-5018 (Part 1) | Upon insertion, 42-day continuous exposure, and removal
  Percent of subjects who are tolerant of TAR-302-5018 indwelling for the designated period of time and do not require TAR-302-5018 removal prior to the scheduled date of removal due to meeting any of the Subject Stopping Criteria or other drug or device constituent related adverse event.
Tolerability of TAR-302-5018 (Part 2) | Upon insertion, 84-day continuous exposure, and removal
  Percent of subjects who are tolerant of TAR-302-5018 indwelling for the designated period of time and do not require TAR-302-5018 removal prior to the scheduled date of removal due to meeting any of the Subject Stopping Criteria or other drug or device constituent related adverse event.
Pharmacokinetic Analysis of Plasma and Urine (Part 1) | From Day 0 to Day 56
  Analysis of plasma trospium exposure and urinary trospium exposure.
Pharmacokinetic Analysis of Plasma and Urine (Part 2) | From Day 0 to Day 112
  Analysis of plasma trospium exposure and urinary trospium exposure.
Reduction in incontinence over baseline (Part 1) | From Day 0 to Day 84
  A negative change from baseline in number of daily episodes of urinary incontinence, where incontinence is defined as an incident of involuntary loss of urine.
Reduction in incontinence over baseline (Part 2) | From Day 0 to Day 112
  A negative change from baseline in number of daily episodes of urinary incontinence, where incontinence is defined as an incident of involuntary loss of urine.
Reduction in daily micturition episodes (Part 1) | From Day 0 to Day 56
  A negative change from baseline in the number of times a subject urinates into the toilet.
Reduction in daily micturition episodes (Part 2) | From Day 0 to Day 112
  A negative change from baseline in the number of times a subject urinates into the toilet.
Increase in voided volume per micturition (Part 1) | From Day 0 to Day 56
  An increase over baseline as measured over separate 24-hour periods.
Increase in voided volume per micturition (Part 2) | From Day 0 to Day 112
  An increase over baseline as measured over separate 24-hour periods.

OTHER OUTCOMES:
Quality of Life (Part 1) | From Day 0 to Day 84
  Evidence of improvement in QoL as assessed by the OAB-q Short Form.
Quality of Life (Part 2) | From Day 0 to Day 112
  Evidence of improvement in QoL as assessed by the OAB-q Short Form.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cutie, MD, Study Director — TARIS Biomedical, Inc.
Locations (12):
- United States (12):
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - DelRicht Clinical Research, LLC, New Orleans, Louisiana
  - Bay State Clinical Trials, Inc, Watertown, Massachusetts
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - New Jersey Urology, Voorhees Township, New Jersey
  - Accumed Research, Garden City, New York
  - Manhattan Medical Resear, New York, New York
  - UWCR - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Urology of Virginia, Virginia Beach, Virginia